CLINICAL TRIAL: NCT03533985
Title: The Effect of Music Therapy on Neonates Diagnosed With Neonatal Abstinence Syndrome: A Pilot Study
Brief Title: Effect of Music Therapy on Infants With Neonatal Abstinence Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Joanne Loewy, Director, Louis Armstrong Center for Music and Medicine at Mount Sinai Beth Israel, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 16-1991; IRB 16-00740 (Other: Icahn School of Medicine at Mount Sinai)
Record Dates: First submitted 2018-05-11; First posted 2018-05-23 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: NAS
Keywords: Neonatal Abstinence Syndrome; Music therapy; Attachment; Music medicine; Multi-modal stimulation
MeSH Terms: conditions — Neonatal Abstinence Syndrome

STUDY DESIGN:
Intervention Model Description: Counterbalancing will be achieved by assigning a different order of presentation of conditions for each group. Participants will remain in the study for two weeks, but continue to receive music therapy for the duration of their stay in the NICU.
Who Masked: Participant, Outcomes Assessor
Masking Description: Parents of infants will be unaware of the interventions' effects. Outcomes Assessor will be unfamiliar with desired outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Song of Kin (Experimental): Voice (with or without guitar)- lullaby/ Holding meter
  Interventions: Behavioral: Song of Kin
- Gato box (Experimental): Simple rhythms using Remo Gato box will be played by the MT-BC using a 3rd to comfort, engage or sedate
  Interventions: Other: Gato box
- Ocean disc (Experimental): Creating a consistent womb-like sound soundscape to comfort, engage or sedate
  Interventions: Other: Ocean disc
- Contingent singing (Experimental): Provision of communicative vocalization-"parantese" to engage with infants, prosodic responses to infant cues (eye contact, body position)
  Interventions: Other: Contingent singing
- Tonal Vocal holding (Experimental): Providing a 'blanket of tone' to comfort, engage or sedate
  Interventions: Other: Tonal Vocal holding
- Muted shaker (Experimental): If infant is awake, the muted shaker will be used to entrain to the infant's vital signs-to comfort, soothe or sedate
  Interventions: Other: Muted shaker

INTERVENTIONS:
Behavioral: Song of Kin — Music therapists will assess meaningful song/theme (of choice/culture) and provide musical elements in a way that nurtures parents. They will then develop a simplified part of the theme into a soothing lullaby for their infants to be utilized directly by the parent/s and/or the music therapist to comfort, engage or sedate.
  Other Names: Music psychotherapy with parent/s
  Arms: Song of Kin
Other: Gato box — Depending on the time of intervention and need of the infant the music therapist will provide rhythmic entrainment that follows the heart rate or suck patterns of the infant
  Other Names: Rhythmic entrainment
  Arms: Gato box
Other: Ocean disc — Depending on the time of intervention and needs of the infant the music therapist will provide a whoosh sound using the Remo Ocean disc. It will be entrained to the infant's respiratory rate.
  Other Names: Timbre entrainment
  Arms: Ocean disc
Other: Contingent singing — Depending on the state of the infant, the music therapist will provide short segments of conversant prosody, to enhance quiet-alert, or stimulate relaxation/sleep
  Arms: Contingent singing
Other: Tonal Vocal holding — Music therapist will provide a vowel, long held tone, sung without vibrato
  Arms: Tonal Vocal holding
Other: Muted shaker — If infant is awake, the muted shaker will be used to entrain to the infant's vital signs-to comfort, soothe or sedate
  Arms: Muted shaker

SUMMARY:
This study examines the effects of 6 different music therapy interventions on outcomes for neonates diagnosed with Neonatal Abstinence Syndrome.

DETAILED DESCRIPTION:
The purpose of this exploratory pilot study is to learn what, if any, effects live music therapy interventions have on the pacification, stabilization, and development of infants diagnosed with Neonatal Abstinence Syndrome (NAS). Neonatal Abstinence Syndrome is a group of problems that occur in a newborn who has been exposed to illegal or prescription opiates while in the mother's womb. Participants will receive 6 music therapy sessions over a 14-day period based on a randomized treatment schedule of 6 different interventions.

ELIGIBILITY:
Inclusion Criteria:

Infants who meet the following inclusion criteria will be eligible to participate in the study irrespective of race, religion, ethnicity, or gender:

* Admitted to the NICU immediately postpartum
* Gestational age 28 weeks or older
* No identified hearing disorder
* Do not have a diagnosed developmental disability (i.e. Down Syndrome)
* Do not have Fetal Alcohol Syndrome
* Medically cleared to participate in the study by nurse or neonatologist
* Parent or legal guardian able/willing to give consent & complete the PBQ (Postpartum Bonding Questionnaire)

Exclusion Criteria:

* Admitted to the NICU at any time other than immediately postpartum
* Gestational age <28 weeks old
* Has an identified hearing disorder
* Has diagnosed developmental disability (i.e. Down syndrome)
* Has Fetal Alcohol Syndrome
* Is not medically cleared to participate in the study by the nurse or neonatologist
* Parent or legal guardian unable/unwilling to give consent

Min Age: 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Heart Rate | up to 2 weeks
Respiratory Rate | up to 2 weeks
O2 sats | up to 2 weeks
  Oxygen saturation levels (O2 sats)
Activity level | up to 2 weeks
  The neonatologist or nurse will assess and mark as active/alert, active to stimulation, flaccid, hypertonic, hypotonic, irritable, jittery, lethargic, paralyzed&medicated, quiet, sedated, or tremors
Sleep category | up to 2 weeks
  The neonatologist or nurse will assess and mark as quiet sleep, active sleep, drowsy state, alert inactivity, fussing or crying.
Feeding (sucking and absorption) category | up to 2 weeks
  The neonatologist or nurse will rate feeding (sucking/absorption) from 1 (active/perpetual) to 12 (none/gavage)
Neonatal Abstinence Scoring (NAS) | up to 2 weeks
  The NAS score lists 21 symptoms that are most frequently observed in opiate-exposed infants. Each symptom and its associated degree of severity are assigned a score and the total abstinence score is determined by totalling the score assigned to each symptom over the scoring period. Please provide the full scale info (example 0 (no symptoms) to 10 (severe symptoms)

SECONDARY OUTCOMES:
Postpartum Bonding Questionnaire (PBQ ) | Baseline
  Questionnaire to assess capacity for attachment in both mothers and fathers. 25 item scale with each item rated from always to never. Scoring is based on four categories: impaired bonding scores 0-60, rejection and pathological anger scores 0-35, infant-focused anxiety scores 0-20, and incipient abuse scores 0-10. Total range from 0 (good bonding) to 125 (poor bonding).

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Loewy, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Kathy Murphy, PhD, Principal Investigator — Loyola University; Aimee Telsey, MD, Study Director — Icahn School of Medicine at Mount Sinai
Locations (6):
- United States (6):
  - Tulane University Hospital, New Orleans, Louisiana
  - Joseph M. Sanzari Children's Hospital, Hackensack, New Jersey
  - Northwell Health, New Hyde Park, New York
  - Mount Sinai West, New York, New York
  - Maria Fareri Children's Hospital, Valhalla, New York
  - Drexel University/Hahnemann Hospital-College of Nursing and Health Professions, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loewy J, Stewart K, Dassler AM, Telsey A, Homel P. The effects of music therapy on vital signs, feeding, and sleep in premature infants. Pediatrics. 2013 May;131(5):902-18. doi: 10.1542/peds.2012-1367. Epub 2013 Apr 15. PMID 23589814
- [Background] Loewy J. NICU music therapy: song of kin as critical lullaby in research and practice. Ann N Y Acad Sci. 2015 Mar;1337:178-85. doi: 10.1111/nyas.12648. PMID 25773633
- [Background] Bieleninik L, Ghetti C, Gold C. Music Therapy for Preterm Infants and Their Parents: A Meta-analysis. Pediatrics. 2016 Sep;138(3):e20160971. doi: 10.1542/peds.2016-0971. Epub 2016 Aug 25. PMID 27561729
- [Derived] Pahl A, Young L, Buus-Frank ME, Marcellus L, Soll R. Non-pharmacological care for opioid withdrawal in newborns. Cochrane Database Syst Rev. 2020 Dec 21;12(12):CD013217. doi: 10.1002/14651858.CD013217.pub2. PMID 33348423
- See also: Related Info — http://nicumusictherapy.com